CLINICAL TRIAL: NCT00707876
Title: A Phase II, Open Label, Randomized, Multicenter Trial Comparing Noncontrast MRA Versus Ferumoxytol Vascular Enhanced MRI (VE-MRI) for the Detection of Clinically Significant Stenosis or Occlusion of the Aortoiliac and Superficial Femoral Arteries in Subjects With Peripheral Arterial Disease Scheduled for Digital Subtraction Angiography (DSA)
Brief Title: Magnetic Resonance Angiography for Peripheral Arterial Disease (PAD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: FER-PAD-001
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Arterial Disease (PAD)
Keywords: Peripheral arterial disease (PAD); Magnetic Resonance Angiography (MRA); Magnetic Resonance Imaging (MRI), imaging agent or biomarker
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Dose 1 versus non-contrast MRA
  Interventions: Drug: ferumoxytol
- 2 (Experimental): Dose 2 versus non-contrast MRA
  Interventions: Drug: ferumoxytol
- 3 (Experimental): Dose 3 versus non-contrast MRA
  Interventions: Drug: ferumoxytol

INTERVENTIONS:
Drug: ferumoxytol — Dose 1 versus non-contrast MRA
  Arms: 1
Drug: ferumoxytol — Dose 2 versus non-contrast MRA
  Arms: 2
Drug: ferumoxytol — Dose 3 versus non-contrast MRA
  Arms: 3

SUMMARY:
The purpose of this study is to compare the difference between two magnetic resonance imaging (MRI) techniques for visualizing arteries. The study hypothesizes that one method that relies upon imaging flowing blood in the pelvic and leg arteries will not be as accurate or efficient as injecting a safe imaging agent to change the appearance of the blood on the MRI. Both methods will be compared with Digital Subtraction Angiography (DSA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with symptoms of PAD
* Scheduled for DSA

Exclusion Criteria:

* Critical leg ischemia manifested by ulcers, gangrene or leg amputation
* Laboratory evidence of iron overload, liver disease, pregnancy
* History of allergy to or recent exposure to radiocontrast, gadolinium chelates, or intravenous iron therapy
* Clinical concerns about co-morbidities, subject suitability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
To assess sensitivity and specificity of non-contrast MRA and VE-MRI at three ferumoxytol dosing levels | 3 weeks

SECONDARY OUTCOMES:
To assess positive and negative predictive values of VE-MRI using ferumoxytol at different dosing levels. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Strauss, MD, Study Director — AMAG Pharmaceuticals, Inc.
Locations (1):
- Lexington, Massachusetts, United States